CLINICAL TRIAL: NCT04447482
Title: A Prospective, Randomized, Multi-center, Superiority Clinical Study to Evaluate the Effectiveness and Safety of Bronchoscopic Lung Biopsy Under the Guide of CT Stereotactic Auxiliary Equipment and Accessories
Brief Title: ENB Vs. Conventional Bronchoscopy With Fluoroscopy for Safe and Effective Biopsy of Pulmonary Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Youhe Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202001131102-CT
Record Dates: First submitted 2020-05-08; First posted 2020-06-25 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Lung Neoplasms; Pulmonary Neoplasm
Keywords: Peripheral Pulmonary Lesion; Lung Biopsy; Electromagnetic Navigation Bronchoscopy; Bronchoscopy; Fluoroscopy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): 4D electromagnetic navigation bronchoscopy (4D-ENB) for lung biopsy. Guidance based on tip tracked surgical tools and images calculated from CT.
  Interventions: Device: ENB with image-guided lung biopsy
- Control Group (Active Comparator): Bronchoscopic lung biopsy taken while using X-ray fluoroscopy.
  Interventions: Procedure: Conventional Bronchoscopy guided by Fluoroscopy

INTERVENTIONS:
Device: ENB with image-guided lung biopsy — Electromagnetic navigational bronchoscopy system with tip tracked instruments.
  Other Names: SPiN Thoracic Navigation System™
  Arms: Treatment Group
Procedure: Conventional Bronchoscopy guided by Fluoroscopy — Bronchoscopic lung biopsy with fluoroscopy.
  Arms: Control Group

SUMMARY:
Evaluate results for participants with lung lesions randomized to either 4D Electromagnetic Navigation Bronchoscopy (4D-ENB) versus Conventional Bronchoscopy with Fluoroscopy for diagnostic biopsy and detection of lung cancer.

DETAILED DESCRIPTION:
The objective of this clinical trial is to evaluate the safety and efficacy results for two bronchoscopic biopsy techniques for sampling lung lesions: either image-guided electromagnetic navigation or conventional bronchoscopy with fluoroscopy. The diagnostic yield and adverse events of participants prospectively randomized to either arm will be evaluated. This is a prospective, randomized, multi-center study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be selected:

  1. Be older than 18 (including 18) and younger than 75 (including 75);
  2. The population with peripheral lung lesions detected in chest CT scanning and who require biopsy;
  3. The subjects are willing to undergo bronchoscopy and meet the requirements for bronchoscopy;
  4. The subjects or their guardians can understand the trial objective, volunteer to participate and sign the informed consent form.

Exclusion Criteria:

* Subjects will be excluded if they meet any of the following criteria:

  1. The patient is participating in another drug or medical device clinical trial (drug clinical trial within 3 months or medical device clinical trial within 1 month);
  2. Women of childbearing age who have positive pregnancy test result and lactating women;
  3. Allergic to anesthetics;
  4. Bronchoscopy contraindications, including: active massive hemoptysis; recent myocardial infarction or unstable angina pectoris; severe heart and lung dysfunction; severe hypertension and arrhythmia; uncorrectable bleeding tendency (such as severe coagulation disorders, uremia and severe pulmonary hypertension); severe superior vena cava obstruction syndrome; suspected aortic aneurysm; multiple pulmonary bullae; systemically extreme exhaustion.
  5. Visible intraluminal lesions found during bronchoscopy;
  6. Patients with severe lung diseases (including: severe bronchodilatation, severe emphysema, etc.) and patients determined to be unsuitable for the examination by the investigators;
  7. Patients with a pacemaker or defibrillator;
  8. Patients who cannot cooperate with the doctor to complete bronchoscopy, such as patients with mental and neurological diseases, mental retardation and mental disorders;
  9. Patients to whom bronchoscopy and bronchoscopic sampling are not applicable to diagnose the lesions, or other patients determined to be unsuitable for this trial by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic rate of lung biopsies between the treatment group and the control group. | 6 months.
  Diagnostic rate is defined as the proportion of true positive and true negative.

SECONDARY OUTCOMES:
Sampling success rate of the treatment group and the control group. | 2 weeks.
  Sampling success rate means the proportion of lung nodules and abnormal lung tissues in all tissues sampled from bronchoscopic lung biopsy.
Navigation time (time to find the lesions) of the treatment group and the control group. | Duration of procedure, or up to 120 minutes.
  For this outcome, duration of procedure is defined as the time from the biopsy tool reaching the main carina (registration) to the biopsy tool reaching the lesion.
Total operation time of the treatment group and the control group. | Duration of procedure, or up to 120 minutes.
  For this outcome, duration of procedure is defined as the time from the bronchoscopy accessing the glottis for the first time to bronchoscopy exiting the glottis for the last time.
Navigation success rate of 4D-ENB and biopsy accessories. | Duration of procedure, or up to 120 minutes.
  Navigation success rate is defined as the proportion of the biopsy tools reaching the lung tissues. For this outcome, duration of procedure is defined as the time from the biopsy tool reaching the main carina (registration) to finishing the biopsy for the last time.
Device performance evaluation of CT Stereotactic Auxiliary Equipment and Accessories. | Duration of procedure, or up to 120 minutes.
  Device performance means the functions, reliability, safety and accessibility of the system. Performance will be evaluated by observing these characteristics during the procedure. For this outcome, duration of procedure is defined as the time from the biopsy tool reaching the main carina (registration) to finishing the biopsy for the last time.

CONTACTS AND LOCATIONS:
Overall Officials: Cathaly Hong, Study Director — Shanghai Youhe Medical Technology Co., Ltd.
Locations (4):
- China (4):
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang
  - Shanghai Changhai Hospital, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Shanghai East Hospital, Shanghai

REFERENCES:
- [Background] Raval AA, Amir L. Community hospital experience using electromagnetic navigation bronchoscopy system integrating tidal volume computed tomography mapping. Lung Cancer Manag. 2016 Apr;5(1):9-19. doi: 10.2217/lmt-2015-0007. Epub 2016 Apr 8. PMID 30643545
- [Background] Flenaugh, E.L., & Mohammed, K.H.. Initial Experience Using 4D Electromagnetic Navigation Bronchoscopy System With Tip Tracked Instruments For Localization of Peripheral Lung Nodules. The Internet Journal of Pulmonary Medicine 18(1): 1-7, 2016.